CLINICAL TRIAL: NCT03091894
Title: Dexmedetomidine Added to Propofol for Drug Induced Sleep Endoscopy in Adult Patients With Obstructive Sleep Apnea: A Prospective Randomized Controlled Trial
Brief Title: Dexmedetomidine Added to Propofol for Drug Induced Sleep Endoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Essam Fathi (Other Government)
Responsible Party: Sponsor-Investigator, Essam Fathi, assistent professor, Zagazig University
Organization: Zagazig University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 3-2017-021
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: Dexmedetomidine; Sleep; Endoscopy; Propofol
MeSH Terms: interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- propofol (Active Comparator): patients will receive only propofol intravenous infusion for sedation
  Interventions: Drug: Propofol
- propofol-dex. (Active Comparator): patients will receive dexmedetomidine in addition to propofol intravenous infusion for sedation
  Interventions: Drug: Propofol; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Propofol — propofol intravenous infusion via syringe pump with loading dose of 0.5 mg/kg over 3 minutes then continuous infusion in a dose of 25-75 ug/kg/minute
  Other Names: diprivan
Drug: Dexmedetomidine — dexmedetomidine intravenous infusion via syringe pump with loading dose of 0.5ug/kg over 5 minutes the continuous infusion in a dose of 0.2-0.7ug/kg/hour in addition to the propofol infusion as in propofol group
  Other Names: precedex
  Arms: propofol-dex.

SUMMARY:
This study evaluate the effect of adding dexmedetomidine intravenous infusion to propofol intravenous infusion during sedation for drug induced sleep endoscopy. Twenty five patients will receive propofol only while the other twenty five will receive propofol and dexmedetomidine.

DETAILED DESCRIPTION:
Propofol is a commonly used intravenous anesthetic drug used for procedural sedation. Dexmedetomidine is an alpha 2 adrenergic receptor agonist which has a sedative and analgesic effects.In the current study the success of the sedation during drug induced sleep endoscopy will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years
* patients with obstructive sleep apnea
* ASA 1and2

Exclusion Criteria:

* patient refusal
* age less than 18 years
* morbid obesity
* known or suspected allergy to the studied drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-09 (Actual); Primary Completion 2018-04-08 (Actual); Study Completion 2018-04-08 (Actual)

PRIMARY OUTCOMES:
success of sedation | the duration of the procedure under sedation is usually about 20 minutes
  to complete the procedure with diagnosis of site and degree of obstruction

SECONDARY OUTCOMES:
time until sufficient sedation | about 5-10 minutes from start of sedation
  time till patient is ready to start endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: essam f abdelgalel, A.professor, Principal Investigator — Zagazig University
Locations (1):
- Zagazig university, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No